CLINICAL TRIAL: NCT05536492
Title: Autologous Fibrin Glue Mixed With Bone Graft(Sticky Bone) and Advanced Platelet Rich Fibrin Compared to Conventional Alveolar Ridge Preservation Technique : Randomized Controlled Trial
Brief Title: Sticky Bone Compared to A-PRF(Platlet Rich Fibrin) Effect on Alveolar Ridge Preservation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arab American University (Palestine) (Other)
Responsible Party: Principal Investigator, Ahmad Nassar, dentist and clinical Msc student, Arab American University (Palestine)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRC/HC/1087/22
Record Dates: First submitted 2022-09-05; First posted 2022-09-13 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: A-PRF; ALLOGRAFT
MeSH Terms: interventions — Transplantation, Homologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- G1-Control group (No Intervention): normal socket healing after extraction without intervention
- G2 (Experimental): SOCKET AUGMENTATION WITH A-PRF ALONE
  Interventions: Procedure: A-PRF
- G3 (Experimental): SOCKET AUGMENTATION WITH A-PRF + ALLOGRAFT
  Interventions: Procedure: A-PRF; Procedure: ALLOGRAFT

INTERVENTIONS:
Procedure: A-PRF — EXTRACTION FOR SINGLE rooted tooth followed by augmentation with PRF
  Arms: G2; G3
Procedure: ALLOGRAFT — EXTRACTION FOR SINGLE rooted tooth followed by augmentation with PRF + ALLOGRAFT
  Arms: G3

SUMMARY:
In this research investigators are going to detect the effect of using different type of materials(sticky bone\platlet rich fibrin ) compared to normal healing on the dimensional changes of alveolar crest after single rooted tooth extraction by using CBCT (cone-beam computed tomography) at time of extraction and after 16-24 weeks

DETAILED DESCRIPTION:
Patients who are treated and referred for having extractions in the upper and lower arch for single rooted teeth will have CBCT for each patient at time of extraction (T0) and after 3 months (T1) , by using the cross sectional of the CBCT investigators will measure the difference from the middle of the socket to buccal and palatal\lingual walls at 3 different points below the crest 1mm, 3mm , 5mm .

* the thickness of the buccal bone at baseline (T0) at 1, 3 and 5 mm below the crest
* the horizontal ridge width at crest- 1 mm (HW- 1 mm), crest- 3 mm (HW- 3 mm) and crest- 5 mm (HW- 5 mm) at the buccal/palatal side, in millimetres and later transformed to percentages
* the vertical resorption on both buccal and palatal side, in millimetres
* the socket fill defined as the highest point of viewable mineralized bone at the middle of the socket; absolute values (in mm) and percentages were calculated by comparing the initial depth of the socket and the depth after three months of healing preparation of the materials to be augmented : autologous fibrin glue mixed with bone graft(sticky bone) would be prepared by using green tubes by choukroun company centrifuged at 1300 rpm for 14 minutes (using DUE centrifuge) then mixed with 0.5 cc FDBA and the exudate of the compressed A-PRF then applied to the extraction site A-PRF PLUGS will be prepared using red tubes using venous blood centrifuged at 1300 rpm for 14 min , then the compressed using special tray and applied in the extraction sockets

ELIGIBILITY:
Inclusion Criteria:

* presence of the buccal and palatal/lingual bony walls evaluated clinically by measuring the thickness of the alveolar ridge and radiologically by a CBCT , and residual periodontal attachment of at least 6 mm of single rooted tooth

Exclusion Criteria:

* complicated tooth extraction, and any medical problem that could interfere with the mucosal and bony healing processes or contraindicating an implant placement, such as anticoagulation, antiaggregatory medication, radiotherapy, bisphosphonate therapy, diabetes, endocarditis risk factors, immunosuppression, and renal or hepatic failure

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
RIDGE DIMENSIONS | 4 Months
  USING CBCT
BONE DENSITY | 4 MONTHS
  USING CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- ArabAmericanU, Ramallah, West Bank, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No